CLINICAL TRIAL: NCT05743660
Title: Key circRNA Identification of Postoperative Delirium in Elderly Patients Undergoing Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: XuzhouCH20220629
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-02

CONDITIONS: Postoperative Delirium
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma is isolated from peripheral blood to extract plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- POD group: According to the occurrence of postoperative delirium, the patients were divided into POD group and non-POD group
- non-POD group: According to the occurrence of postoperative delirium, the patients were divided into POD group and non-POD group

SUMMARY:
The observational study aims to discover differentially expressed circRNAs in the peripheral blood of patients with postoperative delirium, which aims to answer the main questions at:

Whether there are changes in circRNA expression in peripheral blood in elderly patients with delirium after cardiopulmonary bypass surgery? Whether the circRNA with altered expression plays an important role in the occurrence and development of POD? What are the functions and underlying mechanisms of circRNA with altered expression in POD? Voluntary patients will receive follow-up 1 day before and 7 days after surgery to assess their cognitive function, and peripheral blood will be collected 1 day before and 3 days after surgery. The study divided patients into POD group and non-POD group according to whether delirium occurred within 7 days after surgery.

DETAILED DESCRIPTION:
Investigators combined qRT-PCR by performing circRNAs chip analysis to study differential expression of circRNAs in plasma samples of elderly patients with non-POD who underwent cardiac surgery under general anesthesia and cardiopulmonary bypass. Subsequently, miRNA binding sites and associated mRNAs are predicted by bioinformatics analysis. Moreover, we plan to construct predicted circN-MIRNA-MRNA co-expression networks to study the main functions and pathways of target genes, thereby attempting to provide a preliminary view of the potential role of a circRNA in POD. The study may provide an important perspective on the differential expression of circRNA in patients with POD, and may also provide insights into biomarkers and therapeutic targets of POD.

ELIGIBILITY:
Inclusion Criteria:

1. Be over 50 years old;
2. ASA Grade I-III;
3. Heart surgery is planned under general anesthesia.

Exclusion Criteria:

1. Patients with the second surgery;
2. The ejection fraction is less than 40%;
3. The score of the preoperative simple mental status examination (MMSE) is less than 24 points;
4. Patients with mental illness or central nervous system disease;
5. Patients who cannot or refuse to complete MMSE before surgery.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing heart surgery
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Differences in circRNA microarrays before and after surgery | 1 day before surgery，3 day after surgery
  Plasma was isolated from peripheral blood, RNA samples were prepared, and circRNA microarray analysis was performed. The differences in circRNA expression in peripheral blood of POD patients and non-POD patients were comprehensively analyzed.
3-minute Diagnostic Interview for CAM | Consecutive 7 days after the surgery
  Postoperative delirium was assessed by 3-minute Diagnostic Interview for confusion assessment method (CAM).

CONTACTS AND LOCATIONS:
Overall Officials: Yangzi Zhu, Doctor, Principal Investigator — Xuzhou Central Hospital; Liwei Wang, Doctor, Study Director — Xuzhou Central Hospital
Locations (1):
- Xuzhou Central Hospital, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No